CLINICAL TRIAL: NCT00194155
Title: Cytomegalovirus Infection and Pregnancy Outcomes
Brief Title: Cytomegalovirus (CMV) Infection in Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: R01 17625-03-13
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Pregnancy Complications; Cytomegalovirus Infection
Keywords: cytomegalovirus; pregnancy; placenta
MeSH Terms: conditions — Pregnancy Complications; Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Case-Only

SUMMARY:
The purpose of this study is to determine if (recurrent) cytomegalovirus (CMV) infection of the mother results in pregnancy complications such as preterm delivery, severe preeclampsia, poor fetal growth, or stillbirth.

DETAILED DESCRIPTION:
CMV infection in adults with a normal immune system is rarely a serious event. Once a person has been infected with CMV, they may have recurrences (relapses) of the infection. If a mother is infected with the virus or relapses during pregnancy, her fetus may be at risk for infection. Unlike infection in adults, fetal infection may result in serious complications (congenital infection). The effects of fetal infection with CMV are well understood and many efforts have been made to potentially reduce the risk of congenital infection. However, the effect of CMV infection on the pregnancy itself (when the fetus is not affected by CMV) is less understood.

In this study, we plan to determine if CMV recurrence in the mother results in pregnancy complications. The pregnancy complications listed above have been associated with poor placental function. We also plan to determine if (recurrent) CMV infection in the mother is associated with CMV infection of the placenta.

ELIGIBILITY:
Inclusion Criteria:

* Women who deliver at term without pregnancy complications
* Women who deliver (preterm, less than 37 weeks gestation) as a result of spontaneous preterm labor
* Women whose pregnancies are complicated by severe preeclampsia
* Women whose pregnancies are complicated by unexplained poor fetal growth (less than the 10th percentile).
* Women whose pregnancies are complicated by unexplained stillbirth.

Exclusion Criteria:

* Women with multi-gestational pregnancies, or whose pregnancies are complicated by a congenital malformation or chromosomal abnormality.
* Women who have a medical history of hypertension (high blood pressure), diabetes, or severe renal (kidney) disease

Min Age: 15 Weeks | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will use already collected clinical samples in order to test for cytomegalovirus (CMV), in order to determine whether CMV is associated with pregnancy complications that are attributed to placental dysfunction. The subject population will include women diagnosed with preeclampsia, intrauterine fetal demise, intrauterine growth restriction, and spontaneous pre-term delivery. There will also be healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2003-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Parry, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States